CLINICAL TRIAL: NCT06128278
Title: Acute Equol Supplementation and Vascular Function in Postmenopausal Women With and Without CKD
Brief Title: Acute Equol Supplementation and Vascular Function in Women With and Without CKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-0070
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases; Vascular Function; Women
Keywords: S-equol; Chronic Kidney Disease; Vascular Function; Women
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Equol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- (1) S-equol, (2) Placebo (Experimental): This is a randomized, placebo-controlled, crossover study. Participants in one arm will receive S-equol (one visit) and then placebo (the other visit).
  Interventions: Drug: S-equol; Other: Placebo
- (1) Placebo, (2) S-equol (Experimental): This is a randomized, placebo-controlled, crossover study. Participants in one arm will receive placebo (one visit) and then S-equl (the other visit).
  Interventions: Drug: S-equol; Other: Placebo

INTERVENTIONS:
Drug: S-equol — Oral supplementation of S-equol
Other: Placebo — Oral supplementation of placebo

SUMMARY:
The risk of cardiovascular disease (CVD) is significantly elevated in patients with chronic kidney disease (CKD). Notably, women with CKD commonly experience menstrual disturbances induced by CKD, which may contribute to impaired vascular function and elevated CVD risk. However, most of the literature in nephrology focuses on male patients, and studies on women's vascular health are limited. Establishing effective therapies for improving vascular function and reducing CVD risk in women with CKD is a high research priority of the NIH.

Equol contributes to improvement in vascular function, mediated in part by its anti-oxidative and anti-inflammatory properties. However, there is no information on the effect of equol on vascular function in women with CKD. The proposed project aims to determine the acute effect (1-hour, 2-hours, and 3-hours post ingestion) of oral equol supplementation on vascular function in postmenopausal women with and without CKD.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) have a significantly higher risk of cardiovascular diseases (CVD). Indeed, CVD is the leading cause of death in these patients. A primary reason why CKD so greatly exacerbates CVD risk is that CKD accelerates vascular dysfunction, including endothelial dysfunction (i.e., reduced brachial artery flow-mediated dilation [FMDBA]) and increased arterial stiffness (i.e., reduced compliance of the large-elastic arteries such as carotid artery), mediated in part by oxidative stress and inflammation that subsequently reduce the bioavailability of nitric oxide (NO; a vasodilator). Given CKD affects 15% of the U.S. population and 13% of the global population, CKD and its associated CVD risk are major public health concerns.

Women with CKD commonly experience menstrual disturbances, amenorrhea, and/or early menopause. Impaired ovarian function is well-known to compromise vascular health and increase CVD risk even in healthy women. As such, the vasculature of women with CKD may be exposed to the detrimental effects of both CKD and impaired ovarian function, which is secondary to CKD and menopause. Thus, declining kidney function and reduced circulating levels of cardioprotective sex hormones, particularly estradiol (E2), are two interrelated factors that contribute to vascular dysfunction and elevated CVD risk in women with CKD.

The long-term use of hormone replacement therapy (HRT) in postmenopausal women is controversial due to studies reporting its adverse effects on cardiovascular risk and breast cancer, which resulted from the long-term use of HRT. Current guidelines reserve the use of HRT only for short-term treatment of menopausal symptoms (e.g., vasomotor), prevention of bone loss and fractures, hypoestrogenism caused by hypogonadism, surgical menopause, or primary ovarian insufficiency. In women with CKD, limited studies examined the effect of HRT. Given reduced vascular dysfunction (associated with reduced circulating E2 secondary to CKD and menopause) and high CVD risk in postmenopausal women with CKD, there is a strong need for the identification of alternative pharmacological compounds to HRT that can improve vascular function in this population.

Equol is a gut microbiota-derived secondary metabolite of soy isoflavone (i.e., daidzein) and is an estrogen receptor (ER) β agonist. Equol has been identified as a vasoactive nutraceutical and has been shown to benefit vascular function in preclinical studies and clinical studies including healthy subjects. Similar to E2, the beneficial effect of equol on vascular function appears to be in part mediated by its anti-inflammatory and anti-oxidative properties that subsequently increase NO production. However, whether equol improves vascular function in postmenopausal women with CKD is unknown.

The overall goal of the proposed 2-period, double-blind, randomized, placebo-controlled, crossover pilot study is to evaluate the acute effect (1-hour, 2-hours, and 3-hours post-ingestion) of equol supplementation on vascular function (i.e., FMDBA and carotid compliance) and circulating markers of oxidative stress and inflammation in postmenopausal women with and without stage 3-4 CKD. This pilot study will also provide an effect size for designing a future trial testing the chronic effect of equol on vascular function in women with stage 3-4 CKD.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal (50-69 y) women
2. Women with CKD including stage 3-4 (eGFR 15-59 ml/min/1.73m2) determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) 2021 equation
3. Women without CKD (eGFR >60 ml/min/1.73m2) must be healthy (free from hypertension, kidney disease, CVD, diabetes, and other chronic disease as assessed by self-report, medical history, and screening labs).

Exclusion Criteria:

1. Use of HRT or has used HRT for <6 months prior to enrollment
2. Advanced CKD requiring dialysis
3. History of kidney transplant
4. Use of immunosuppressant medications (unless taking a stable dosage for a quiescent disease)
5. Current tobacco or nicotine use or history of use in the last 12 months
6. Antioxidant and/or omega-3 fatty acid use within the 2 weeks prior to testing
7. Marijuana use within 2 weeks prior to testing
8. Consumption of soy and soy-based products 3 days prior to testing
9. Uncontrolled hypertension in CKD group (BP>140/90 mmHg)
10. Atrial fibrillation
11. Active infection or antibiotic therapy
12. Hospitalization in the last month

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Brachial Artery Flow-Mediated Dilation | Baseline; 1-hour, 2-hours, and 3-hours post ingestion
  Flow-mediated dilation of the brachial artery will be performed using ultrasonography and analyzed with a commercially available software package as percent change in diameter from baseline following reactive hyperemia.

SECONDARY OUTCOMES:
Change in Carotid Femoral Pulse Wave Velocity | Baseline; 2-hour post ingestion
  A transcutaneous custom tonometer [Noninvasive Hemodynamics Workstation (NIHem), Cardiovascular Engineering Inc.] will be used to non-invasively assess carotid femoral pulse wave velocity.
Change in oxidative stress markers | Baseline; 1-hour, 2-hours, and 3-hours post ingestion
  8-isoprostane
Change in inflammation markers | Baseline; 1-hour, 2-hours, and 3-hours post ingestion
  interleukin-6, tumor necrosis factor-α
Change in S-equol concentrations | Baseline; 1-hour, 2-hours, and 3-hours post ingestion
  Plasma S-equol levels

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in CKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).